CLINICAL TRIAL: NCT05805800
Title: Olanzapine and 5-HT3 With or Without Dexamethasone to Prevent Nausea and Vomiting Induced by Chemotherapy: A Non-inferiority, Prospective, Multi-Centered, Randomized, Controlled, Phase III Clinical Trial
Brief Title: Olanzapine and 5-HT3 With or Without Dexamethasone to Prevent CINV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xingchen Peng (Other)
Responsible Party: Sponsor-Investigator, Xingchen Peng, Ph.D,Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-157
Record Dates: First submitted 2023-03-27; First posted 2023-04-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5HT3RA+Olanzapine (Experimental): Using one of the 5-HT3 receptor antagonists within 30 minutes before cisplatin/adriamycin/cyclophosphamide.On day 1-4, Olanzapine is delivered orally after dinner.
  Interventions: Drug: 5HT3RA+Olanzapine
- 5HT3RA+Olanzapine+Dexamethasone (Active Comparator): Using one of the 5-HT3 receptor antagonists within 30 minutes before cisplatin/adriamycin/cyclophosphamide.On day 1-4, Olanzapine is delivered orally after dinner.On first day, dexamethasone is given orally within 30 minutes before cisplatin/adriamycin/cyclophosphamide administered.
  Interventions: Drug: 5HT3RA+Olanzapine+Dexamethasone

INTERVENTIONS:
Drug: 5HT3RA+Olanzapine — Using one of the 5-HT3 receptor antagonists within 30 minutes before cisplatin/adriamycin/cyclophosphamide.
  On day 1-4, Olanzapine is delivered orally after dinner.
  Arms: 5HT3RA+Olanzapine
Drug: 5HT3RA+Olanzapine+Dexamethasone — Using one of the 5-HT3 receptor antagonists within 30 minutes before cisplatin/adriamycin/cyclophosphamide.
  On day 1-4, Olanzapine is delivered orally after dinner. On first day, dexamethasone is given orally within 30 minutes before cisplatin/adriamycin/cyclophosphamide administered.
  Arms: 5HT3RA+Olanzapine+Dexamethasone

SUMMARY:
Nausea and vomiting caused by chemotherapy are considered by patients as the main side effects of cancer treatment, which affect the quality of treatment and life.At present, NCCN guidelines have recommended three or four drug regimens for highly emetic chemotherapy (HEC) to prevent vomiting, all containing dexamethasone.However, its side effects such as moderate to severe insomnia, hyperglycemia, dyspepsia, upper abdominal discomfort, irritability, increased appetite, weight gain and acne are gathering increasing concerns.For certain patients, the use of dexamethasone should be avoided.Analysis shows that olanzapine can replace the effect of dexamethasone.Hence, the investigators initiated this prospective, multi-center, phase III study to validate the dexamethasone-free protocol: removing dexamethasone from a three drug regimen containing olanzapine, dexamethasone, and 5-HT3RA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older with malignant disease；
2. Life expectancy ≥ 3 months;
3. Scheduled to receive highly emetogenic chemotherapy；
4. Had a European Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Exclusion Criteria:

1. There are contraindications to chemotherapy(Absolute number of neutrophils ≤ 1,500/uL, hemoglobin ≤ 90g/L, platelet count ≤ 10000/uL, serum creatinine level ≥ 2.0mg/dl (177 μmol/L), ALT and AST ≥ 2.5 times the upper normal limit, bilirubin ≥ 1.5 times the upper normal limit);
2. History of central nervous system disease (e.g., brain metastases or a seizure disorder);
3. Severe cognitive impairment；
4. Treatment with another antipsychotic agent such as risperidone, quetiapine, clozapine, a phenothiazine, or a butyrophenone within 30 days before enrollment or plans for such treatment during the study period;
5. Concurrent use of pharyngeal or abdominal radiotherapy;
6. Concurrent use of quinolone antibiotics;
7. Concurrent use of Amifostine;
8. Chronic alcoholism;
9. Known hypersensitivity to olanzapine;
10. Know arrhythmia, uncontrolled congestive heart failure or acute myocardial infarction within 6 months;
11. Known uncontrolled diabetes mellitus;
12. Vomiting or retching 24 hours before chemotherapy;
13. Use of anti-emesis drugs 48 hours before chemotherapy;
14. Patients who require medication with dexamethasone for pretreatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
0-120h Complete Remission Rate | 24 hours ,48 hours, 72 hours, 96 hours, 120 hours after chemotherapy
  The ratio of patients who have no vomiting and apply no anti-nausea drugs during the whole observation period.

SECONDARY OUTCOMES:
25-120 hours Complete Remission Rate | 24 hours ,48 hours, 72 hours, 96 hours, 120 hours after chemotherapy
  The ratio of patients who have no vomiting and apply no anti-nausea drugs during the 25-120 hours observation period.
0-120h No Nausea Rate | 24 hours, 48 hours, 72 hours, 96 hours, 120 hours after chemotherapy
  The ratio of patients who have no nausea during the whole observation period.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng TL, Hutton B, Clemons M. Chemotherapy-Induced Nausea and Vomiting: Time for More Emphasis on Nausea? Oncologist. 2015 Jun;20(6):576-83. doi: 10.1634/theoncologist.2014-0438. Epub 2015 May 6. PMID 25948677
- [Background] Yang LQ, Sun XC, Qin SK, Cheng Y, Shi JH, Chen ZD, Wang QM, Zhang HL, Hu B, Liu B, Zhang QY, Wu Q, Wang D, Shu YQ, Dong J, Han BH, Wang KM, Dang CX, Li JL, Wang HB, Li BL, Lu JG, Zhang ZH, Chen YX. Efficacy and safety of fosaprepitant in the prevention of nausea and vomiting following highly emetogenic chemotherapy in Chinese people: A randomized, double-blind, phase III study. Eur J Cancer Care (Engl). 2017 Nov;26(6):e12668. doi: 10.1111/ecc.12668. Epub 2017 Apr 10. PMID 28393417
- [Background] Hu Z, Cheng Y, Zhang H, Zhou C, Han B, Zhang Y, Huang C, Chang J, Song X, Liang J, Liang H, Bai C, Yu S, Chen J, Wang J, Pan H, Chitkara DK, Hille DA, Zhang L. Aprepitant triple therapy for the prevention of chemotherapy-induced nausea and vomiting following high-dose cisplatin in Chinese patients: a randomized, double-blind, placebo-controlled phase III trial. Support Care Cancer. 2014 Apr;22(4):979-87. doi: 10.1007/s00520-013-2043-9. Epub 2013 Nov 26. PMID 24276953
- [Background] Tan L, Liu J, Liu X, Chen J, Yan Z, Yang H, Zhang D. Clinical research of Olanzapine for prevention of chemotherapy-induced nausea and vomiting. J Exp Clin Cancer Res. 2009 Sep 23;28(1):131. doi: 10.1186/1756-9966-28-131. PMID 19775450
- [Background] Navari RM, Qin R, Ruddy KJ, Liu H, Powell SF, Bajaj M, Dietrich L, Biggs D, Lafky JM, Loprinzi CL. Olanzapine for the Prevention of Chemotherapy-Induced Nausea and Vomiting. N Engl J Med. 2016 Jul 14;375(2):134-42. doi: 10.1056/NEJMoa1515725. PMID 27410922
- [Background] Chelkeba L, Gidey K, Mamo A, Yohannes B, Matso T, Melaku T. Olanzapine for chemotherapy-induced nausea and vomiting: systematic review and meta-analysis. Pharm Pract (Granada). 2017 Jan-Mar;15(1):877. doi: 10.18549/PharmPract.2017.01.877. Epub 2017 Mar 15. PMID 28503222
- [Derived] Chen S, Pei YY, Zhang HW, Chen Y, Deng LC, Chen X, Wei ZG, Li D, Li ZH, Li RD, Liu ZR, Peng XC. Randomized, double-blind phase III trial of a dexamethasone-free regimen for managing highly emetogenic chemotherapy-induced nausea and vomiting. Int J Cancer. 2026 Jan 1;158(1):131-139. doi: 10.1002/ijc.70069. Epub 2025 Jul 30. PMID 40735921